CLINICAL TRIAL: NCT01864837
Title: Availability of Tongue Diagnosis System for Assessing Tongue Coating Thickness of Patients With Functional Dyspepsia: Study Protocol for Comparative Trial With Conventional Method
Brief Title: Evaluation on the Availability of Tongue Diagnosis System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jin-sung Kim, Full professor, Korea Health Industry Development Institute
Other Study IDs: KOMCIRB-2013-01
Record Dates: First submitted 2013-05-22; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Tongue Coating Thickness
Keywords: tongue coating thickness; tongue diagnosis system; tongue coating percentage; availability; diagnostic device

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Functional dyspepsia: They should meet the Rome III criteria for functional dyspepsia.

SUMMARY:
The aim of the proposed study is to investigate the agreement between the measurement of the tongue diagnosis system (TDS) and the conventional way of tongue diagnosis about the tongue coating thickness (TCT) in the tongue diagnosis of the traditional Korean medicine (TKM).

DETAILED DESCRIPTION:
Tongue diagnosis is one of the important diagnostic techniques to examine the physiologic functions and pathologic changes of the internal organs in TKM.

However, traditional tongue diagnosis has inevitable limitations because of the clinician's subjectivity and environmental factors influencing on the diagnostic results.

Therefore, it is necessary to investigate the availability of the tongue diagnosis system (TDS).

The aim of the this study is to investigate the agreement between the measurement of TDS and the conventional way of tongue diagnosis about TCT in the tongue diagnosis of TKM. So, we will assess the agreement between the measurement of TDS and the final diagnosis of 5 clinicians with five or more years of clinical experience about TCT.

Additionally, we will evaluate the reproducibility of TDS. In the 2nd visit, taking tongue images of each patient with TDS will be performed again at 30 minute-intervals in the same way. And then, we will compare the two TDS measurements of each patient about TCT.

After twice examination of TDS, the weight of tongue coating (mg) will be measured quantitatively by tongue scraping to analyze the correlation between the weight of tongue coating and the measurements of TDS.

In addition, after the collection of 60 patients' tongue images is completed, we will ascertain the validity of the five clinicians for diagnosing the TCT by assessing the inter-and intra-rater reliability of the five clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older
* One who meet the Rome III criteria for functional dyspepsia
* One who is able to read, write, hear, see something
* One who agree on consent form

Exclusion Criteria:

* Mental disorders
* Pregnancy
* Severe systemic organ diseases such as cancer
* Infectious or other serious consumptive diseases
* Geographic tongue
* One who cannot open his/her mouth or protrude his/her tongue

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with functional dyspepsia which be considered to appear the various aspects of tongue coating in traditional Korean medicine(TKM).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
tongue coating thickness(TCT) by tongue diagnosis system | 2nd visit (1st visit is for screening)
  In the 2nd visit, Tongue coating thickness(TCT) will be assessed by tongue coating percentage(%)from TDS measurements. In the advanced study, 29.06% is a cut-off point to separate no coating and thin coating, and 63.51% is a cut-off point to separate thin coating and thick coating.

SECONDARY OUTCOMES:
tongue coating thickness(TCT) by the five clinicians | After completing the collection of 60 patients' tongue images
  After the collection of 60 patients' tongue images is completed, 5 clinicians with five or more years of clinical experience will assess the TCT of 60 patients with 60 images obtained by TDS. In order to decide the final diagnosis of the 5 clinicians as a gold standard, if we have a disagreement among them, we will agree to the views of the majority.
the weight of tongue coating | 2nd visit (1st visit is for screening)
  The weight of tongue coating (mg); It will be measured quantitatively to analyze the correlation between the tongue coating percentage measured with TDS and the weight of tongue coating obtained by tongue scraping(Yaegaki's method).

CONTACTS AND LOCATIONS:
Overall Officials: Jinsung Kim Kim, doctorate, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Korean Medicine Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Son J, Jang S, Nam DH, Han G, Yeo I, Ko SJ, Park JW, Ryu B, Kim J. Availability of tongue diagnosis system for assessing tongue coating thickness in patients with functional dyspepsia. Evid Based Complement Alternat Med. 2013;2013:348272. doi: 10.1155/2013/348272. Epub 2013 Sep 15. PMID 24159343